CLINICAL TRIAL: NCT06960369
Title: Efficacy of Repeated Transcranial Magnetic Stimulation Combined With a Live Probiotic Tablet (Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus Cereus Tablets, Live) in Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Soochow University (Other)
Responsible Party: Principal Investigator, Rui Li, Chief of the Department of Gastroenterology, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024518
Record Dates: First submitted 2025-04-19; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Irritable Bowel Syndrome; Irritable Bowel Syndrome With Diarrhea (IBS-D); Repetitive Transcranial Magnetic Stimulation (rTMS); Probiotic; Chronic Diarrhea; Intestinal Flora
Keywords: Irritable Bowel Syndrome with diarrhea (IBS-D); Repetitive Transcranial Magnetic Stimulation (rTMS); Probiotic
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- rTMS combined with Live Probiotic tablet (Experimental): rTMS combined with Live Probiotic tablet (Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus cereus Tablets, Live).
  rTMS group received 1 Hz/s, 20 min for 2 week; Live Probiotic tablet group received tablets orally, 150 mg three times a day for 2 week.
  Interventions: Combination Product: rTMS combined with Live Probiotic tablet
- rTMS combined placebo (Experimental): rTMS combined placebo
  rTMS group received 1 Hz/s, 20 min for 2 week; placebo group received tablets orally, 150 mg three times a day for 2 week.
  Interventions: Device: rTMS combined placebo
- shamrTMS combined with Live Probiotic tablet (Experimental): shamrTMS combined with Live Probiotic tablet(Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus cereus Tablets, Live)
  Live Probiotic tablet group received tablets orally, 150 mg three times a day for 2 week, shamrTMS group received 0 Hz/s, 20 min for 2 week.
  Interventions: Drug: shamrTMS combined with Live Probiotic tablet
- shamrTMS combined placebo group (Other): shamrTMS combined placebo group
  shamrTMS group received 0 Hz/s, 20 min for 2 week; placebo group received tablets orally, 150 mg three times a day for 2 week.
  Interventions: Other: shamrTMS combined placebo group

INTERVENTIONS:
Combination Product: rTMS combined with Live Probiotic tablet — rTMS group received 1 Hz/s, 20 min for 2 week; Live Probiotic tablet group received tablets orally, 150 mg three times a day for 2 week.
  Arms: rTMS combined with Live Probiotic tablet
Device: rTMS combined placebo — rTMS group received 1 Hz/s, 20 min for 2 week; placebo group received tablets orally, 150 mg three times a day for 2 week.
  Arms: rTMS combined placebo
Drug: shamrTMS combined with Live Probiotic tablet — Live Probiotic tablet group received tablets orally, 150 mg three times a day for 2 week, shamrTMS group received 0 Hz/s, 20 min for 2 week.
  Arms: shamrTMS combined with Live Probiotic tablet
Other: shamrTMS combined placebo group — shamrTMS group received 0 Hz/s, 20 min for 2 week; placebo group received tablets orally, 150 mg three times a day for 2 week.
  Arms: shamrTMS combined placebo group

SUMMARY:
To evaluate the overall efficacy of repeated Transcranial Magnetic Stimulation(rTMS) combined with a Live Probiotic tablet (Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus cereus Tablets, Live) in Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)

Methods:

Clinical efficacy evaluation of TMS combined with Live Probiotic tablet for chronic diarrhea in IBS patients. The 400 IBS patients who meet the recruitment criteria for the clinical study will be randomized into 100 patients in rTMS combined with Live Probiotic tablet (Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus cereus Tablets, Live), rTMS combined placebo, shamrTMS combined with Live Probiotic tablet(Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus cereus Tablets, Live) and shamrTMS combined placebo group. Corresponding treatment was given for 2 week, rTMS group received 1 Hz/s, 20 min for 2 week; Live Probiotic tablet group received tablets orally, 150 mg three times a day for 2 week, shamrTMS group received 0 Hz/s, 20 min for 2 week; placebo group received tablets orally, 150 mg three times a day for 2 week. Clinical assessment included symptoms, stool traits, mood, and sleep.

2. Study on the mechanism of using intestinal flora data to evaluate the treatment of chronic diarrhea in IBS patients. 30 cases each were included in the 4 groups of IBS-eligible patients, and repeated transcranial magnetic stimulation treatment was given to the patient group for 2 week, and the patient group underwent the assessment of investigating the quantity and metabolic changes of the intestinal flora in feces before and after the treatment.

DETAILED DESCRIPTION:
A large number of literature has reported that repetitive transcranial magnetic stimulation(rTMS) can relieve chronic pain. The specific mechanisms include that rTMS can change the excitability of the cerebral cortex, improve cerebral blood flow and metabolism, regulate neurotransmitter and gene expression, and plastic changes in the nervous system.Previous research results revealed that the neural circuit of the cuticular nucleus - anterior cingulate cortex is a unique neural circuit regulating chronic visceral pain in the IBS animal model. To explore the improvement of chronic visceral pain sensitivity in patients with irritable bowel syndrome (IBS) by Transcranial magnetic stimulation (TMS). On this basis, To further explore whether repetitive transcranial magnetic stimulation can treat the diarrhea symptoms of patients with irritable bowel syndrome, and to provide a more reliable and effective treatment method for clinical application.

Objective:

To evaluate the overall efficacy of repeated Transcranial Magnetic Stimulation(rTMS) Combined with a Live Probiotic tablet (Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus cereus Tablets, Live) in Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D), including abdominal diarrhea symptoms,bowel symptoms, and psychiatric symptoms (anxiety, depression, sleep disturbance). And also to explore the mechanism of rTMS combined with Live Probiotic tablet for the treatment of IBS-D, based on intestinal flora data.

Methods:

Clinical efficacy evaluation of TMS combined with Live Probiotic tablet for chronic diarrhea in IBS patients. The 400 IBS patients who meet the recruitment criteria for the clinical study will be randomized into 100 patients in rTMS combined with Live Probiotic tablet (Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus cereus Tablets, Live), rTMS combined placebo, shamrTMS combined with Live Probiotic tablet(Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus cereus Tablets, Live) and shamrTMS combined placebo group. Corresponding treatment was given for 2 week, rTMS group received 1 Hz/s, 20 min for 2 week; Live Probiotic tablet group received tablets orally, 150 mg three times a day for 2 week, shamrTMS group received 0 Hz/s, 20 min for 2 week; placebo group received tablets orally, 150 mg three times a day for 2 week. Clinical assessment included symptoms, stool traits, mood, and sleep.

2. Study on the mechanism of using intestinal flora data to evaluate the treatment of chronic diarrhea in IBS patients. 30 cases each were included in the 4 groups of IBS-eligible patients, and repeated transcranial magnetic stimulation treatment was given to the patient group for 2 week, and the patient group underwent the assessment of investigating the quantity and metabolic changes of the intestinal flora in feces before and after the treatment.

The intestinal flora data of the four groups were analyzed to compare the differences between the treatment groups and control group before and after treatment and the improvement values of the clinical observation indexes were correlated.

ELIGIBILITY:
Inclusion Criteria:

1. Must meet the diagnostic criteria for Irritable Bowel Syndrome of Rome IV.
2. Age range between 18-70 years.
3. The duration of the disease is more than 6 months.
4. There are no pathologic abnormalities or biochemical changes that could explain the bowel-related symptoms.
5. The IBS symptom severity score at baseline must not be less than 75.
6. No pharmacological treatment (excluding emergency treatment) for IBS for at least 2 weeks prior to the start of treatment; no concurrent participation in other clinical programs.
7. Voluntarily sign the relevant informed consent form and voluntarily participate in this clinical project.

Exclusion Criteria:

1. Be less than 18 years old or more than 70 years old.
2. Those who suffer from severe liver, kidney, hematopoietic system diseases, cardiovascular and cerebrovascular diseases, and psychiatric diseases that significantly affect cognitive function.
3. Patients with clear organic diseases of the intestinal tract; patients with diabetes, hyperthyroidism and other systemic diseases that affect the digestive tract dynamics; patients who have had a history of surgery on the anus and intestines or the abdomen.
4. The presence of the following conditions affecting the efficacy or safety judgment: ① regular use of preparations and drugs affecting gastrointestinal dynamics or function; ② treatment with other treatments and drugs that may affect the results of the judgment.
5. Those who are pregnant, breastfeeding or less than 12 months after delivery.
6. Patients with severe fear of needles, metal allergies or sensitivities, or those with pacemakers.
7. Patients who do not comply with the randomized assignment to the treatment group or have a tendency to be unstable such as poor compliance.
8. Patients who are participating in other research projects.
9. Those who do not want to sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of defecation and Bristol Stool Form Scale score | One day before treatment, the first day after the end of treatment, and follow-up until the third month after treatment
  The therapeutic effect was evaluated by recording the frequency of defecation and the state of feces of the patients before and after treatment.
  The Bristol Stool Form Scale is to standardize the classification of stool consistency and form.
  * Types 1-2: Hard, lumpy stools (associated with constipation).
  * Types 3-4: Loose or smooth stools (ideal consistency).
  * Types 5-7: Watery, mushy, or liquid stools (linked to diarrhea). The Bristol Stool Form Scale (BSFS) is for monitoring treatment responses to interventions.

SECONDARY OUTCOMES:
IBS-symptom severity score | One day before treatment, the first day after the end of treatment, and follow-up until the third month after treatment
  The criteria were based on the IBS Symptom Severity Score (IBS-SSS), a hierarchical efficacy assessment method.The IBS-SSS consists of five entries assessing the degree of abdominal pain and discomfort, frequency of abdominal pain episodes, the degree of abdominal distension and discomfort, the degree of satisfaction with bowel habits and behaviors, and the degree of impact of intestinal symptoms on life,with a total score of 500 points. A score of 75-175 is considered mild, 176-300 is moderate, and over 300 is severe. Cure was defined as a total IBS symptom severity of less than 75; efficacy was defined as 2-level improvement in total score(e.g., symptoms improved from severe to mild); validity was defined as a 1-level improvement in tatal(e.g., symptoms improved from severe to moderate or symptoms from moderate to mild); and invalidity was defined as no improvement or deterioration in total score.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Li, Principal Investigator — Rui Li Study Principal Investigator The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
This clinical research protocol is just beginning to be studied at this time and sharing is not recommended at this time.